CLINICAL TRIAL: NCT07130825
Title: The Effect of Different Physical Activity Strategy on Cognitive Efficiency and Mental Fatigue Resistance During a Simulated Mental Working Day
Brief Title: The Effect of Different Physical Activity Strategy on Cognitive Efficiency and Mental Fatigue Resistance
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lithuanian Sports University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: LithuananianSportsU-23
Record Dates: First submitted 2025-04-03; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Healthy Adults

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control (Experimental): Healthy young subjects will participate in research "control" condition attending 8 h simulated working day. During simulated working day subjects will perform cognitive tasks (ANAM4, version 4; Vista Life Science, Norman, OK, USA) for 8 times (1 session 11 tests about 45 min). The effect of a mental workday on cognitive function indicators will be evaluated. Same participants will participate in 3 research trials (control, aerobic activity and combined work model).
  Interventions: Other: 8 hours simulated mental workday
- Aerobic activity (Experimental): Healthy young subjects will participate in research "aerobic activity" condition attending 8 h simulated working day. Subjects will cycle 30 min on a veloergometer in a 50 % of maximal capacity before the cognitive tasks and after them (before and after simulated 8 h workday). During simulated working day subjects will perform cognitive tasks (ANAM4, version 4; Vista Life Science, Norman, OK, USA) for 8 times (1 session 11 tests about 45 min).
  The effect of a moderate-intensity aerobic physical activity before and after 8 hours of a mental workday will be evaluated. Same participants will participate in 3 research trials (control, aerobic activity and combined work model).
  Interventions: Other: 8 hours simulated mental workday; Other: Moderate intensity aerobic activity
- Combined work model (Experimental): Healthy young subjects will participate in research "combined work model" condition attending 8 h simulated working day. Subjects will perform cognitive tasks applying combined work model, which means that participants will be changing their positions from sitting on a balance ball to standing while performing cognitive tasks. During simulated working day subjects will perform cognitive tasks (ANAM4, version 4; Vista Life Science, Norman, OK, USA). The effect of a the combined work model on cognitive functions indicators during a simulated 8 h mental working day will be evaluated. Same participants will participate in 3 research trials (control, aerobic activity and combined work model).
  Interventions: Other: 8 hours simulated mental workday; Other: Combined work model

INTERVENTIONS:
Other: 8 hours simulated mental workday — During a simulated 8-hour mental work day, subjects will complete a set of cognitive tests (ANAM4, version 4; Vista Life Science, Norman, OK, USA) 8 times (1 session approximately 45 minutes), with a break of approximately 10 minutes after each session.
Other: Moderate intensity aerobic activity — In one of the conditions, subjects will perform moderate intensity aerobic activity (cycle veloergometer) for 30 min before 8 hours simulated mental workday and after.
  Arms: Aerobic activity
Other: Combined work model — In one of the conditions, subjects will perform cognitive test during 8 hours simulated mental workday applying combined work model (they will work standing and sitting on a balance ball).
  Arms: Combined work model

SUMMARY:
The main aim of this biomedical study is to determine the effect of moderate-intensity aerobic exercise, before and after an 8-hour workday and a combined work model, on the performance and efficiency of cognitive functions during mental work.

There are lack of previous studies analysing the effects of different physical activity strategies on cognitive efficiency and investigating mental fatigue resistance. Limited research in this area shows that the mechanism of the effect of physical activity on mental fatigue resistance is still unclear. This research will aim to investigate different physical activity strategies, such as combined work model and moderate intensity physical activity before and after office workday, and their impact on a mental and emotional fatigue, cognitive efficiency, sympathetic and parasympathetic systems and metabolic indicators during mentally demanding 8 h workday.

DETAILED DESCRIPTION:
Prolonged sedentary behavior and sustained cognitive workload during typical office workdays contribute significantly to the onset of acute mental fatigue (Kunasegaran et al., 2023). This condition is linked to physiological mechanisms such as reduced cerebral blood flow, diminished glucose availability and transport to active brain regions (García et al., 2021; Kennedy & Scholey, 2000), as well as hormonal alterations (Miyashita & Williams, 2006; Wiehler et al., 2022). These changes negatively impact cognitive efficiency, motivation, and overall brain function (Kunasegaran et al., 2023; Tran et al., 2020). While existing evidence supports the positive influence of physical activity on physical and mental health (Calderwood et al., 2021; Jacquet et al., 2021), there remains a lack of research specifically examining how different physical activity strategies influence cognitive efficiency and resistance to mental fatigue.

This study aims to address this gap by investigating the effects of various physical activity interventions, including a combined work-exercise model and moderate-intensity aerobic exercise performed either before or after an 8-hour mentally demanding workday. Outcomes will focus on mental and emotional fatigue, cognitive efficiency, autonomic nervous system activity (sympathetic and parasympathetic balance), and metabolic responses. By evaluating these parameters, the study seeks to clarify the potential of targeted physical activity strategies to enhance mental fatigue resistance and support cognitive performance in occupational settings. The findings are expected to contribute valuable insight into the development of effective workplace interventions that promote employee well-being, productivity, and resilience.

ELIGIBILITY:
Inclusion Criteria:

* BMI from 18.5 to 24.9 kg/ m2;
* No chronic non-communicable diseases;
* No mental illnesses or disorders;
* No cancer and no chemotherapy in the last 5 years;
* No hearing impairment;
* No smoking;
* No psychotropic substances;
* Heart rate (HR) about 60 bpm at rest;
* Unimpaired color vision;
* Unimpaired or corrected vision;
* Systolic blood pressure from 90 to 139 mmHg, and diastolic - from 50 to 89 mmHg at rest.

Exclusion Criteria:

* mental, oncological, metabolic, cardiovascular, skeletal, muscular, respiratory system disorders or diseases, impaired color vision.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2031-03-01 (Estimated); Study Completion 2031-03-01 (Estimated)

PRIMARY OUTCOMES:
Body mass and body composition (kg) | 2 times in the mornings (day 1 and day 2) of each 3 conditions.
  Body mass and composition (in kilograms) will be evaluated using Tanita Body Composition Analyzer (Japan).
Height (m) | 2 times in the mornings (day 1 and day 2) of each 3 conditions.
  Height (in meters) will be measured using a Harpenden anthropometer set (Holtain Ltd, UK).
Brain hemodynamic response | Before, immediately after the simulated mental workday, 3 hours after the simulated mental workday, and 12 hours recovery after a simulated mental workday in 3 conditions.
  To measure and evaluate hemodynamic response, a functional near-infrared (fNIRS) device NIRx NIRS Sport2 (Medical Technologies LLC-NIR-Scout, USA) with 8 near-infrared (NIR) radiation sources and 7 photodetectors will be used. The photodetectors record the relative changes in oxygen and oxygenated hemoglobin at 7.81 Hz for both wavelengths. The probes are placed at the manufacturer's specified locations to capture the hemodynamic response of the prefrontal cortex. Live recording will be monitored for 6 minutes.
Cognitive performance | Day 1 in 3 different conditions, in 1 condition 8 times for 45 minutes.
  Automated Neuropsychological Assessment Metrics Test Set (ANAM4, version 4; Vista Life Science, Norman, OK, USA). 11 tests will be selected, reflecting the three main cognitive functions - memory, attention and executive function. 11 tests: Procedural RT, Memory search, Spatial processing simultaneous, Matching grids, Matching to sample, Stroop colour word test, Code substitution-learning and Code substitution-delayed, Running memory continuous performance, Continous performance test - traditional. To assess cognitive performance, during a simulated 8-hour mental work day, the subjects will complete a set of cognitive tests 8 times (1 session approximately 45 minutes), after each session there will be a break of approximately 10 minutes. Participants were familiarized with the test battery twice before the experiments.
Blood pressure (mmHg) | 11 times during 1 condition (total 33 times).
  Systolic and diastolic blood pressure (in mmHg) will be measured using a blood pressure monitor (Biolight, Patient Monitor S10, Guangdong Biolight Meditech Co, Hamburg, Germany).
Heart rate and heart rate variability (ms) | During 1 condition rest measurements in the morning, during brain hemodynamic response (3 times during 1 condition), during every session of 8 hours simultaneous mental work day, total 3 conditions.
  Heart rate (HR) will be recorded using a heart rate monitor (Polar H10, Kempele, Finland) with an electrode strap around the chest throughout the study. 5-min RR interval file will then be analyzed using Kubios HR Variability Analysis Software 2.0 (Biomedical Signal and Medical Image Analysis Group, Department of Applied Physics, University of Kuopio, Kuopio, Finland).
Glucose level (mmol/l) | 9 times during 1 condition (total 27 times).
  Glucose level will be measured from capillary blood using Akray glucose analyzer (CONTOUR®PLUS ELITE; Basel, Switzerland). Capillary blood samples will be taken by a qualified medical professional (general practice nurse) at the LSU Institute of Sports Science and Innovation laboratory.
Ketones level (mmol/L) | 9 times during 1 condition (total 27 times).
  Ketones level will be measured from capillary blood using a ketone analyzer (The On Call® GK Dual; San Diego, CA; USA). Capillary blood samples will be taken by a qualified medical professional (general practice nurse) at the LSU Institute of Sports Science and Innovation laboratory.
Lactate level (mmol/L) | 9 times during 1 condition (total 27 times).
  Lactate levels will be measured using a lactate analyzer (Lactatte Pro 2, Arkray, Koji Konan-cho, Koka-shi, Japan). Capillary blood samples will be taken by a qualified medical professional (general practice nurse) at the LSU Institute of Sports Science and Innovation laboratory.
Salivary cortisol concentration (µg/dl) | 11 times during 1 condition (total 33 times).
  The saliva samples will be collected to measure cortisol level (in µg/dl) using an ELISA kits and a Spark multimode microplate reader (Tecan, Austria).
Salivary testosterone concentration (µg/dl) | 11 times during 1 condition (total 33 times).
  The saliva samples will be collected to measure cortisol level (in µg/dl) using an ELISA kits and a Spark multimode microplate reader (Tecan, Austria).
Salivary female sex hormones concentration (pgmol/L) | 11 times during 1 condition (total 33 times).
  The saliva samples will be collected to measure cortisol level (in µg/dl) using an ELISA kits and a Spark multimode microplate reader (Tecan, Austria).
Biochemical urine analysis | 2 times during 1 condition (total 6 times).
  The urine sample will be analyzed in the laboratory using a urine analyzer (PocketChem UA, PU-4010, Arkray, Koji, Konan-cho, Koka-shi, Japan). The analyzer will determine the concentrations of ketones.
Pupil diameter (mm) | Before and 3 times during simulated 8 hours workday in 1 condition (total 12 times).
  The dilation and contraction of the pupils of the test subjects' eyes will be recorded using a special camera (Gazepoint, Vancouver, Canada), which will be placed under the computer screen, in front of the subject.
The psycho-emotional state: Dundee Stress State Questionnaire (DSSQ) | Before and 8 times during simulated 8 hours workday in 1 condition (total 27 times).
  The psycho-emotional state of the subjects will be assessed using the Dundee Stress State Questionnaire (DSSQ). The DSSQ questionnaire will be used to assess the subjects' motivation in relation to the content of the task, performing a cognitive test battery during the mental work day. 15 questions will be used, e.g.: "the content of the task was interesting", "I wanted to do the task well compared to others", etc. The subject will have to mark the corresponding answers to each question, where 4 (strongly), 3 (very), 2 (a little), 1 (a little), 0 (not at all).
The psycho-emotional state: the VAS scale | Before and 8 times during simulated 8 hours workday in 1 condition (total 27 times).
  Motivation, mental fatigue and mind wondering will be assessed using a visual analogue scale (VAS). Subjects will mark their feelings on a 10 centimetres horizontal line from 0 ("completely unmotivated"; "not mentally tired"; "no mind wandering") to 100 ("maximum motivated"; "maximum mental fatigue"; "maximum mind wandering").
The psycho-emotional state: Stanford sleepiness scale. | Before and 8 times during simulated 8 hours workday in 1 condition (total 27 times).
  The Stanford Sleepiness Scale will be used to assess subjects' sleepiness. On this scale, subjects will mark their level of sleepiness from 1 "I feel active, efficient, lively, alert or awake" to 7 "I can no longer fight sleep, I will fall asleep quickly; thoughts are like dreams".
Measurement of maximal aerobic capacity | Before.
  The maximal aerobic capacity of the subjects will be measured in order to determine the average aerobic load, which will be applied in the study condition "aerobic activity ". The subjects will perform a consistently increasing load until complete fatigue on a bicycle ergometer (Lode B.V., Excalibur Sport, Groningen, Netherlands). Throughout the test, subjects will have their heart rate monitored using a chest strap heart rate monitor (Polar H10, Kempele, Finland). A spirometry system (Metalyzer 3B, Cortex, Leipzig, Germany) will be used to measure oxygen uptake (VO2). VO2max (maximum oxygen uptake) will be considered the highest oxygen uptake during any 15 s of exercise.
Sleep quality assessment | 3 days before each condition and during testings.
  Sleep (hours of total sleep and sleep stages) will be monitored using a Garmin wrist-worn watch (Vivo fit 4, UK).
Physical activity assessment | 3 days before each condition and during testings.
  Physical activity (steps per day) will be monitored using a Garmin wrist-worn watch (Vivo fit 4, UK).
Biochemical urine analysis | 2 times during 1 condition (total 6 times).
  The urine sample will be analyzed in the laboratory using a urine analyzer (PocketChem UA, PU-4010, Arkray, Koji, Konan-cho, Koka-shi, Japan). The analyzer will determine the concentrations of leukocytes.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Sport Science and Innovations, Kaunas, Lithuania